CLINICAL TRIAL: NCT00697424
Title: Investigation of Methods to Detect Respiratory Irregularities in Obstructive Sleep Apnea (OSA)
Brief Title: Comparison of Breathing Events Detected by the SleepStyle 200 Auto Continuous Positive Airway Pressure (CPAP) Device to Attended Polysomnography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Jessica Hayward, Fisher & Paykel Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FPHHC254a; AKY/03/07/166
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All subjects will be placed on continuous positive airway pressure (CPAP) therapy during a full night sleep study or polysomnography (PSG). The subjects will spend 2 hours on sub-therapeutic CPAP 4 cmH2O of pressure and the remainder on there therapeutic pressure. Values reported on the device will be compared to scored values from manual scoring of the sleep study.
  Interventions: Device: SleepStyle 200 Auto Series CPAP Humidifier

INTERVENTIONS:
Device: SleepStyle 200 Auto Series CPAP Humidifier — The device will record on internal software perceived sleep disordered breathing events. Events will also be scored manually on the polysomnography (PSG. Results will then be compared.

SUMMARY:
Obstructive Sleep Apnoea (OSA) is a common sleep-breathing disorder affecting around 2-4% of the population and is characterised by loud snoring, periodic collapse of the upper airway particular to sleep, sleep fragmentation, and sometimes daytime sleepiness. Health consequences include impaired cognitive functioning, quality of life, mood, and increased cardiovascular disease risk. Epidemiological studies have demonstrated that increased morbidity and mortality in a dose response manner with increasing severity of sleep disordered breathing.

The standard treatment for OSA is nasal Continuous Positive Airway Pressure (CPAP), which consists of pressurized air applied to the nose via a mask. Generally a single, optimal pressure is prescribed for a patient based on a full night or partial night study during which the pressure is adjusted by a technician until all sleep disordered breathing (SDB) events are abolished. Despite therapy efficacy, compliance to CPAP therapy is sub-optimal.

Due to low compliance it has become common for healthcare providers to follow up subject therapy efficacy through reporting software inherent in many current CPAP devices. Healthcare providers can use this reported data to make appropriate treatment decisions. For this reason the data needs to be accurate. The SleepStyle™ 200 Auto Series CPAP humidifier is an auto adjusting CPAP which stores comprehensive compliance data. The aim of this study is to compare the reliability of the SleepStyle™ 200 Auto Series CPAP data to laboratory-based PSG in detecting sleep disordered breathing.

Hypothesis: The SleepStyle™ 200 Auto Series reporting features accurately detects indices of sleep disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* Apnea Hypopnea Index (AHI) >15 from diagnostic night
* ≥18 years of age

Exclusion Criteria:

* Contraindicated for CPAP use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | At the end of the sleep study.

SECONDARY OUTCOMES:
Respiratory Disturbance Index (RDI) | At the end of the sleep study (PSG)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Hayward, Msc, Principal Investigator — Fisher & Paykel Healthcare
Locations (1):
- Auckland Hospital, Adult Sleep & Ventilation Service, Auckland City Hospital, Auckland, New Zealand

REFERENCES:
- See also: Sponsors web site — http://www.fphcare.co.nz/